CLINICAL TRIAL: NCT04746001
Title: Artificial Intelligence in the Diagnosis of Orthopaedic Conditions, Particularly Bone Tumours and Infection
Acronym: AIortho
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Collaborators: Keele University (Other)
Responsible Party: Sponsor
Other Study IDs: 281854_47208_2021
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Bone Tumours; Bone Infection; Prosthetic Joint Infection; Prosthetic Infection
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Histological slides and limited sequencing data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection
  Interventions: Diagnostic Test: Genomic sequencing; Diagnostic Test: Histological examination
- Tumours
  Interventions: Diagnostic Test: Genomic sequencing; Diagnostic Test: Histological examination

INTERVENTIONS:
Diagnostic Test: Genomic sequencing — Sequencing data
Diagnostic Test: Histological examination — Images for deep learning

SUMMARY:
Translational research aimed at improving diagnostic accuracy of musculoskeletal infection and musculoskeletal tumours using machine learning applied to clinical data, histopathological sections and genomic sequencing.

ELIGIBILITY:
Inclusion Criteria:

Suspected infection of bone tumour and biopsy taken for analysis

Exclusion Criteria:

Patient doesn't consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected orthopaedic infection (including prosthetic joint infection) or bone tumours
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Sequencing data and identification | 3 years
  Identification of infection and tumours using sequencing data
Histological slides and identification | 3 years
  Deep learning using histological images

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Trust, Oswestry, Shropsire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data may be made available as part of publication